CLINICAL TRIAL: NCT07116642
Title: Comparison of Patient Reported and Clinical Outcome Measures Based on Scar Placement in Patients Undergoing Breast Conserving Surgery (PROM-S Study)
Brief Title: Comparing Patient Reported Outcomes and Clinical Outcomes Based on Different Scar Placement in Patients Undergoing Standard Breast Conserving Surgery for Breast Cancer: The PROM-S Study.
Acronym: PROM-S
Status: Recruiting | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CO24/163189
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer - Female; Surgery of Breast Cancer
Keywords: breast cancer; surgery; patient reported outcomes
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is for patients with breast cancer and the objective is to compare patient reported outcome measures (PROMs) based on scar placement in patients undergoing standard breast-conserving surgery (sBCS). BCS has become the standard of care for eligible patients with breast cancer (current UK national BCS rate is 60%).

Scar placement for sBCS can be divided into two groups: those directly over the cancer, or those in remote locations (e.g. around the nipple, near the armpit, the lower part of the breast, where the breast and the chest meet etc.) with the aim of hiding the scar in more visually acceptable locations on the breast. Multiple factors determine where the scar is placed such as aesthetics, other health conditions, location of the cancer, etc. However, it is currently unclear whether the location of scar placement for sBCS affects patient reported outcomes.

The growing importance on breast cosmesis has led to more attention from clinicians and patients with regards to the selection of surgical incision placement for sBCS. By using a validated questionnaire (BREAST-Q), we wish to assess if there is any difference in PROMs based on scar placement (over the lesion vs. remote) in patients undergoing sBCS.

It is anticipated that the study results will help champion and guide care for future breast cancer patients, as well as providing an insight into how patient satisfaction may vary between different sBCS approaches.

This questionnaire study will include consecutive patients undergoing sBCS at Leeds Teaching Hospitals NHS Trust.

Participation in this non-randomised study will not impact on routine clinical care or decision making for the type of surgery planned or scar placement choice. Patients will be asked to complete the BREAST-Q questionnaire prior to surgery, after 2 weeks, as well as 3 and 12 months after surgery.

DETAILED DESCRIPTION:
Advances in surgical techniques, has led to a growing importance on breast appearance (cosmesis). Presently, scar placement for standard breast conserving surgery (sBCS) can vary from either directly over the cancer or be in remote locations with the aim of hiding the scar in more aesthetically acceptable locations on the breast.

A number of factors dictate the outcome of scar placement such as aesthetics, comorbidities, location of the cancer, etc. However, it is currently unclear whether the location of scar placement for sBCS affects patient reported outcomes in short- or long- term post-surgery as we do not have sufficient information from the patient's point of view of their experience and satisfaction.

We will use a validated patient outcomes questionnaire for breast surgery (BREAST-Q) to compare patient satisfaction with scar placement (over the lesion vs. remote) for patients undergoing sBCS. We hope that the results will provide valuable additional information when future patients are counselled with regards to scar placement.

The principle research objective is to assess the impact of scar placement location on patient reported and clinical outcomes utilising the BREAST-Q questionnaire in patients undergoing standard breast conserving surgery (sBCS).

Secondary objectives include:

* comparing aesthetic outcome (appearance) and functional outcome of standard breast conserving surgery based on scar placement using Patient Reported Outcome Measures (PROMs) from the patients' point of view.
* comparing clinical outcomes between over the lesion vs. remote scar placement in patients undergoing standard breast conserving surgery
* explore potential factors that influence the locations of scar placement for standard breast conserving surgery (surgeon / clinical factors).
* explore the extent of patient involvement in decision-making process This is a single-centre, non-randomised observational study that aims to recruit a minimum of 75 participants. The surgery could be for invasive or non-invasive breast cancer, with or without axilla surgery. All patients will be invited to complete the BREAST-Q patient reported outcome questionnaire on four occasions. The four time points are: before surgery, 2 weeks after surgery and at 3 and 12 months after surgery.The BREAST-Q is a standardised and validated questionnaire that covers symptoms and issues such as physical, sexual and psychosocial well-being, satisfaction with breasts, the impact of radiotherapy and satisfaction with the treating medical team and the level of information provided.

The patient will receive instructions for completing the questionnaires from the study team. These can be completed either in paper forms or electronically. Additionally, socio-demographic and routine clinical data collected as part of standard care (including but not limited to complications and other treatments required, such as radiotherapy) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥18 years of age
* Able to provide written informed consent
* Invasive breast cancer or ductal carcinoma in situ (DCIS) suitable for sBCS (including multifocal cancers requiring x2 wires or magseeds)
* Able to understand and complete the questionnaire

Scar over the lesion defined as radial, transverse, vertical, oblique scar over the tumour lesion location in the breast Remote incisions defined as lateral perimeter/periareolar/infra-mammary fold/ benelli/hemi-batwing

* No restrictions on tumour size (decision on suitability for sBCS will be based on clinical assessment)
* Any axillary nodal staging status
* Bilateral cancers allowed
* Post neo-adjuvant chemotherapy (NACT) allowed

Exclusion Criteria:

* Male patients (BCS not proven as standard of care) or transgender
* Patients undergoing oBCS (such as wise pattern, vertical scar mastopexy incision pattern or volume replacement chest wall perforator flap)
* Patients undergoing mastectomy with or without immediate autologous or implant reconstruction
* Patients requiring nipple excision (central wide local excision)
* Patients undergoing wide local excision under local anaesthetic
* Women not able or willing to give informed consent
* Where close tumour proximity to skin or skin involvement necessitates skin excision over the tumour
* Patients diagnosed with locoregional recurrence
* Patients diagnosed with associated distant metastasis
* Patients undergoing diagnostic excision surgery for atypical breast lesions or benign lesions
* Patients diagnosed with phyllodes lesion
* Patients who have had previous ipsilateral breast surgery (any type)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: Breast cancer patients been treated with surgery at a single site in Leeds, UK
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The BREAST-Q - Breast Conserving Therapy Module | from enrolment to 12 months
  The BREAST-Q is a validated PROM that has been developed for the use in a breast cancer population (Pusic et al. 2009). It can be used to assess the PROMs at pre-operative baseline and at multiple time points after surgery.
  In particular, the Breast Conserving Therapy Module is able to assess multiple domains including physical, sexual and psychosocial well-being, satisfaction with breasts, the impact of radiotherapy and satisfaction with the treating medical team and level of information provided (Klassen et al. 2020). The module uses an independent Rasch 'scales' with overarching themes of psychosocial and physical quality of life. The scores are converted to a Rasch scale 0-100 with higher scores meaning better satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Dr Hartup, PhD, RN, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (1):
- St James's University Hospital, Leeds, West Yorkshire, United Kingdom